CLINICAL TRIAL: NCT02854904
Title: Immune Effect of Dexmedetomidine as Immunomodulatory Anesthesic Agent in Patients Undergoing to Spinal Fusion: a Double-blind, Randomized and Placebo-controlled Clinical Trial
Brief Title: Immune Effect of Dexmedetomidine in Patients Undergoing to Spinal Fusion
Acronym: eMUNODEX
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sarah Network of Rehabilitation Hospitals (Other)
Collaborators: University of Brasilia (Other)
Responsible Party: Principal Investigator, Luciano Pereira Miranda, MD, Sarah Network of Rehabilitation Hospitals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRH1
Record Dates: First submitted 2016-07-26; First posted 2016-08-04 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2016-08

CONDITIONS: Spine; Arthrosis; Spondylolysis; Spondylolysis, Multiple Sites in Spine; Spondylolisthesis
Keywords: Immunomodulatory; dexmedetomidine; anesthesia; alpha-2 agonist; arthrodesis; spinal fusion; Immune effect; double randomized clinical trials
MeSH Terms: conditions — Osteoarthritis; Spondylolysis; Spondylolisthesis; Ankylosis | interventions — Adrenergic alpha-2 Receptor Agonists; Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexmedetomidine intervention (Experimental): Dexmedetomidine (1 ug/kg/hr) during anesthesia.
  Interventions: Drug: Dexmedetomidine intervention
- Placebo (Placebo Comparator): Infusion of normal saline during anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine intervention — Immune effect of alpha-2 agonist to arthrodesis. Dexmedetomidine as a immune control anesthesic in patients undergoing to arthrodesis. Alpha-2 agonist to general anaesthesia.
  Other Names: Alpha-2 agonist; Precedex
  Arms: Dexmedetomidine intervention
Drug: Placebo — Placebo controlled
  Other Names: Comparator
  Arms: Placebo

SUMMARY:
Alpha-agonist in anesthesia display immunomodulatory effect in addition to antiadrenergic control. This effect of the immune system can be a key to a better perioperative safety and quality.

The association of dexmedetomidine at general anesthesia adds up organic protection and inflammatory control to a surgery trauma owing to antinociception and immunomodulatory effect.

The aim this study is evaluate if the association of dexmedetomidine at general anesthesia standing effective immunomodulatory control to trauma and improve changes at outcomes in patients undergoing to spinal fusion.

DETAILED DESCRIPTION:
PURPOSE

Interactions between the hypothalamus-pituitary-adrenal axis, sympathetic nervous system and immunological system acts in the initiation and propagation to reactions of trauma distress. A large number of factors affect the activation of immune response owing to surgical trauma and anesthesia. Regarding the current field, surveys are need to evaluate the real clinical significance of immune control.

In order to blunt the surgical stress response, the control of inflammatory response is considered by many authors the most important factor. Therefore, dexmedetomidine as an immunomodulatory anesthesic agent plays a way to more effective control to the endocrine metabolic response, predicate role to better outcomes in patients undergoing to major surgical trauma.

This trial is designed as a double-blind, randomized and placebo-controlled to evaluate the utility of dexmedetomidine as immunomodulatory anesthetic agent in a major surgical model.

HYPOTHESIS

Dexmedetomidine provide more effective immune control at general anesthesia in patients undergoing to spine fusion.

OBJECTIVES

Goals standard to immune control, hemodynamic safety and recovery quality.

1. Measure of release pro-inflammatory cytokines [interleukin 1-beta (IL-1b), interleukin 6 (IL-6) and tumoral necrosis factor alpha (TNF-a)] to evaluate the anti-inflammatory activity in vivo of dexmedetomidine;
2. Serum dosage of interferon-gamma and interleukin 4 (IL-4) to evaluate changes of cellular and humoral T-helper cells activity;
3. Endocrine-metabolic changes will be evaluated with the dosage serum cortisol, insulin and glucose;
4. Hemodynamic safety will be performed with a vital signals and changes of ventricular stress and myocardium ischemia markers [brain natriuretic pro-peptide (pro-BNP), troponin I and creatine kinase (CK-MB)];
5. Renal function will be evaluated with measure diuresis rate, fluid balance, serum levels of Cystatin-C, electrolytes [sodium and potassium] and arterial blood gas;
6. Time to open eyes after turn off anesthesic gases to evaluate the wake-up time (time to recovery of consciousness (ROC);
7. Partial pressure of carbon dioxide (CO2) and respiratory rate immediately after the end of anesthesia to evaluate a respiratory changes;
8. Ricker Sedation-Agitated Scale and Visual Analogic Pain Scale will be performed after 15 minutes on arrival of patients at the recovery room;
9. The QoR-40 (quality of recovery - 40) questionnaire before the surgery and the first postoperative day to a quality support;
10. The incidence of nausea, vomiting, hypotension, hypertension, bleeding, bradycardia and tachycardia will be recorded during surgery and in a pos anesthetic period.

RESEARCH METHOD

A randomized double-blind clinical trial was elaborated to compare two groups of patients, active dexmedetomidine group (Dexmedetomidine group - SD) and placebo comparator (Placebo group - SP). For our knowledge, our proposal study was approved by the Ethnic Committee of the Sarah Network of Rehabilitation Hospitals since June of 2016 (Approval Number: 50057415.0.0000.0022). All patients who will be enrolled to our study must sign informed consent.

Once schedule spinal fusion, patients both sex, 18 to 75 years old and physical state (ASA) 1-3 will be enrolled in this trial. All patients will be evaluated in the anesthesic ambulatory. Then, the patients will be randomly divided blindly into Group SD or Group SP.

In the pre-anesthesic room, patients will be monitored with electrocardiography, non invasive blood pressure, pulse oximetry and entropy. After peripheral venous access obtained, the first sample (Time 0: Before induction of anesthesia) can be taken and start dexmedetomidine or placebo dripping.

According to a clinic demand, anesthesia will be performed with propofol, rocuronium, fentanyl, methadone and/or remifentanyl. After endotracheal access, the lungs will be ventilated with oxygen in air (1:2), and the ventilation rate will be adjusted to maintain the end-tidal carbon dioxide partial pressure between 35 and 45 mmHg. The concentrations of sevoflurane will be adjusted for maintain hypnosis entropy score between 40 and 45.

Invasive blood pressure through radial artery will be obtained. The samples of blood will be retrieved from arterial line at three moments: Time 1: 8h after the end of surgery; Time 2: 7:00h AM, 24h after the first sample have been collected, and; Time 3: 7:00h AM, 48h after the first sample have been collected.

In the SD group, dripping of dexmedetomidine (0.2 - 1 ug/kg/hr) will be administered during surgery. Already in the SP group, normal saline will be administered with same rate as a placebo.

Effective site concentration of anesthesics drugs will be adjusted for maintain entropy between 40 and 45 and changes of vital sign between 20% of baseline value. On line sevoflurane concentrations using an infrared anesthetic gases analyzer.

After the end of surgery, all anesthetics agents will be discontinued and the time to wake-up will be recorded. Patients will be asked to open their eyes and the time of eyes open will be recorded. After the eyes open, the patients will be transferred to recovery room.

After arrival on the recovery room, blood pressure, heart rate, Ricker Sedation-Agitated Scale and Visual Analogic Pain Scale will be measure in the first 15 minutes and in the leave of recovery room. The time of staying in postanesthetic care unit is recorded.

The incidence of nausea, vomiting, hypotension, hypertension, bleeding, bradycardia and tachycardia will be recorded during surgery and staying at postanesthetic care unit. All participants will be followed for the duration of surgery and postanesthetic period.

STATISTICAL ANALYSIS

All data will be expressed as mean ± standard deviation or absolute values. The Student's t-test or Mann-Whitney U-test to performed to demographic data.

The Wilcoxon rank-sun test to compare cytokines concentrations and scores of quality between groups at the time points. Friedman's test will be performed to compare cytokine or clinical markers among each time points groups. Dunn's pos hoc test for statistic significance.

Recovery and quality profiles [time to recovery of consciousness (ROC); Ricker sedation-agitated scale at the postanesthetic care unit and; QoR-40] will be analyzed by paired t-test.

The incidence of nausea/vomiting, hypotension, hypertension, bleeding, bradycardia, and tachycardia will be analyzed by Chi-square test.

All analyses will be performed using SPSS version 15.0 software for Windows. A P-value < 0.05 will be deemed to a statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III;
* Age > 18;
* Elective surgery to spinal fusion, and;
* Informed consent signed.

Exclusion Criteria:

* Patients with severe heart disease with New York Heart Association class > III;
* Severe arrhythmia;
* Uncontrolled hypertension or hypotension;
* Hemodynamic unstably;
* Hypersensitivity with drugs;
* Cognitive deficiency, dementia, or delirium;
* Weight up to 100 kg and/or body mass index (BMI) greater than or equal to 40;
* Illicit drugs users and/or alcoholic;
* Steroids and/or non-steroids anti-inflammatory chronic users;
* Tricyclic antidepressants users;
* Hepatic or renal compromised and;
* Infective disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2016-08; Primary Completion 2016-11 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline of anti-inflammatory activity | Time 0: 7:00 AM, after obtained peripheral venous access; Time 1: 8h after the end of surgery; Time 2: 7:00h AM, 24h after the first sample have been collected; Time 3: 7:00h AM, 48h after the first sample have been collected
  Measure of release pro-inflammatory cytokines [interleukin 1-beta (IL-1b), interleukin 6 (IL-6) and tumoral necrosis factor alpha (TNF-a)]
Changes from baseline of cellular and humoral T-helper cells activity | Time 0: 7:00 AM, after obtained peripheral venous access; Time 1: 8h after the end of surgery; Time 2: 7:00h AM, 24h after the first sample have been collected; Time 3: 7:00h AM, 48h after the first sample have been collected
  Serum dosage of interferon-gamma and interleukin 4 (IL-4)
The endocrine-metabolic changes | Time 0: 7:00 AM, after obtained peripheral venous access; Time 1: 8h after the end of surgery; Time 2: 7:00h AM, 24h after the first sample have been collected; Time 3: 7:00h AM, 48h after the first sample have been collected
  Serum dosage of cortisol, insulin and glucose

CONTACTS AND LOCATIONS:
Overall Officials: Luciano P Miranda, Principal Investigator — Sarah Network of Rehabilitation Hospitals
Locations (1):
- Luciano Pereira Miranda, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: Undecided
Cause the study not yet start.